CLINICAL TRIAL: NCT00432640
Title: Complete Echo-Endoscopic Staging of Lung Cancer vs Surgical Staging: a Randomized Clinical Trial
Brief Title: Assessment of Surgical sTaging vs Endoscopic Ultrasound in Lung Cancer: a Randomized Clinical Trial (ASTER Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Kurt Tournoy, MD, PhD, University Hospital Ghent
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006/461
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: (suspected) Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Endoscopic ultrasound staging
  Interventions: Procedure: Endoscopic ultrasound staging
- 2 (Active Comparator): Surgical staging
  Interventions: Procedure: Surgical staging

INTERVENTIONS:
Procedure: Endoscopic ultrasound staging — Endoscopic ultrasound staging with both EUS-FNA and EBUS-TBNA
  Arms: 1
Procedure: Surgical staging — Surgical staging
  Arms: 2

SUMMARY:
Lung cancer is one of the most prevalent cancers and has a very high mortality. Both treatment and prognosis depend on the staging. Surgical staging of the mediastinum mainly by means of a cervical mediastinoscopy is the gold standard. Mediastinal staging is however a field that undergoes a fast technological development. Transesophageal ultrasound guided fine-needled aspiration (EUS-FNA) and an endobronchial ultrasound guided transbronchial fine-needled aspiration (EBUS-TBNA) are two complementary endoscopic ultrasound techniques which together allow cytological analysis of all mediastinal lymph nodes. This means that the combination of both techniques enables a complete (bilateral) mediastinal investigation (N2 and N3, except para-aortal station 6).

Hypothesis: complete endoscopic ultrasound staging identifies more patients with locally advanced disease compared to surgical staging (current standard of care).

Study design: A randomized controlled multi-center double arm diagnostic phase III trial, in which patients are randomly assigned to either surgical staging (arm B) or endoscopic ultrasound staging with both EUS-FNA and EBUS-TBNA (arm A).

Arm A: Examination by EUS-FNA and EBUS-TBNA. These techniques are performed in an outpatient one session setting under conscious sedation and take together about 30 to 60 minutes. If no metastasis are shown, the patient undergoes a surgical staging procedure (for confirmation). For reasons of convenience and patient-comfort, the EUS-FNA investigation is performed before the EBUS-TBNA.

Arm B: Surgical staging with either cervical mediastinoscopy, parasternal mediastinoscopy, thorascopic mediastinal exploration or exploratory thoracotomy, performed according to institutional practice.

Patients in whom no lymph node metastasis are found proceed to thoracotomy with systematic lymph node sampling to obtain an accurate intraoperative mediastinal staging.

Primary outcome: The assessment of N2-N3 lymph node metastases.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with NSCLC or with a clinical suspicion for lung cancer in whom mediastinal lymph node invasion (either N2 or N3) is suspected based on the available thoracic imaging
* Pending the results of the mediastinal staging, the patient is otherwise considered a candidate for a surgical treatment with the intention to cure (this is a resectable tumor)
* The patient is clinically fit for diagnostic surgery (this is an operable patient)
* No distant metastasis after routine clinical work up
* Provision of a written informed consent

Exclusion Criteria:

* Former therapy (chemotherapy or radiotherapy or surgery) for lung cancer
* Reasons because of which the patient is unable to swallow the EUS-instrument (e.g. Zenker Divertikel, unexplained esophageal stenosis) or because of which the patient is unable to undergo a bronchoscopy
* Patients who, based on available thoracic imaging, are unlikely to be staged accurately by any surgical staging procedure (mediastinoscopy/ - tomy, VATS)
* Respiratory insufficiency or other contra-indications for bronchoscopy
* Concurrent other malignancies
* Uncorrected coagulopathy
* Study cannot be discussed with the patient (e.g. mental disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
We hypothesize that the combination of EUS and EBUS in an out-patient one-session setting is more sensitive for the detection of locally advanced disease (N2/N3) compared to surgical staging (standard of care)

SECONDARY OUTCOMES:
Assessment of mediastinal tumour invasion (T4)
Assessment of the rate of avoided surgical procedures (arm A)
Assessment of the negative predictive value
Assessment of the difference in the cost for lymph node staging
Assessment of the complication rates
Assessment of the rate of futile thoracotomies
Assessment of quality of life (EQ5D)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Tournoy, MD, PhD, Principal Investigator — University Hospital, Ghent; Jouke Annema, MD, Principal Investigator — Leidens Universitair Medisch Centrum
Locations (4):
- Belgium (2):
  - University Hospital Ghent, Ghent
  - Leuven University Hospital, Leuven
- Leidens Universitair Medisch Centrum (LUMC), Leiden, Netherlands
- Papworth University Hospital, Cambridge, United Kingdom

REFERENCES:
- [Derived] Rintoul RC, Glover MJ, Jackson C, Hughes V, Tournoy KG, Dooms C, Annema JT, Sharples LD. Cost effectiveness of endosonography versus surgical staging in potentially resectable lung cancer: a health economics analysis of the ASTER trial from a European perspective. Thorax. 2014 Jul;69(7):679-81. doi: 10.1136/thoraxjnl-2013-204374. Epub 2013 Sep 24. PMID 24064440
- [Derived] Annema JT, van Meerbeeck JP, Rintoul RC, Dooms C, Deschepper E, Dekkers OM, De Leyn P, Braun J, Carroll NR, Praet M, de Ryck F, Vansteenkiste J, Vermassen F, Versteegh MI, Veselic M, Nicholson AG, Rabe KF, Tournoy KG. Mediastinoscopy vs endosonography for mediastinal nodal staging of lung cancer: a randomized trial. JAMA. 2010 Nov 24;304(20):2245-52. doi: 10.1001/jama.2010.1705. PMID 21098770
- See also: Website of the University Hospital Ghent — http://www.uzgent.be